CLINICAL TRIAL: NCT06502782
Title: Areal and Linear Comparison of the Effect of Gingival Phenotype on Gingival Recession
Brief Title: Areal and Linear Comparison of Gingival Recession
Acronym: agr
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Tuğba ŞAHİN, Assistant professor, Abant Izzet Baysal University
Other Study IDs: 2022/288
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Gingival Recession
Keywords: Gingiva; Gingival recession; Screening
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Thin phenotype: A thickness of 1 mm or less is classified as thin gingival tissue.
  Interventions: Diagnostic Test: digital assesment
- Thick phenotype: A thickness of more than 1 mm is classified as thick gingival tissue.
  Interventions: Diagnostic Test: digital assesment

INTERVENTIONS:
Diagnostic Test: digital assesment — Gingival recession sites were scanned with an intraoral optical surface scanner, and STL images were recorded. The images were imported into image analysis software. The depth, width and area of gingival recession were calculated using Autocat program.

SUMMARY:
Recent advances in digital technology have led to the emergence of precise methods for measuring gingival recession and tissue thickness. This study aimed to compare digital measurement methods and conventional periodontal probe measurements for the assessment of gingival recession influenced by the gingival phenotype.

This study involved 128 gingival recession sites from 28 systemically healthy patients aged 18-45 years. The participants were categorized into two groups on the basis of gingival thickness. The plaque index, gingival index, probing depth, clinical attachment level, gingival recession depth, and gingival recession width, and keratinized gingival thickness and width were measured using a manual periodontal probe and an intraoral optical surface scanner. Statistical analysis was performed with nonparametric tests because the data were not normally distributed. P<0.05 indicated statistical significanct.

ELIGIBILITY:
Inclusion Criteria: The study included systemically healthy subjects aged 18-45 years with systemic disease or systemic disease under control.

Exclusion Criteria: The exclusion criteria were as follows:

* Patients with a history of radiotherapy,
* Patients with chemotherapy,
* Immunosuppressive use,
* Tobacco use,
* Smoking,
* Patients with labially exposed teeth and teeth with prominent root protrusions,
* Pregnancy and lactation,
* Patients with uncontrolled diabetes,
* Patients with postorthodontic extractions,
* Patients with gingival recession, .Patients with gingival enlargement caused by piercing and nail-biting habits.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study included 128 gingival recessions at 128 sites in 28 systemically healthy patients aged 18-45 years old. The patients were divided into two groups according to the thickness of the gingiva in the teeth with gingival recession.
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2022-11-12 (Actual); Primary Completion 2023-11-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
keratinized gingival thickness | Baseline
  Keratinized gingival thickness refers to the vertical measurement of the gingival tissue that extends from the free gingival margin to the mucogingival junction, characterized by a keratinized epithelial layer which provides enhanced protection and stability to the underlying periodontal structures.
keratinized gingival width | Baseline
  Keratinized gingival width refers to the horizontal dimension of the gingival tissue that is keratinized, measured from the free gingival margin to the mucogingival junction.
Gingival recession depth | Baseline
  Gingival recession is the apical migration of the gingival margin away from the cemento-enamel junction (CEJ), resulting in the exposure of the root surface of a tooth.
Gingival recession width | Baseline
  Gingival recession width refers to the horizontal measurement from the exposed cemento-enamel junction (CEJ) to the apical point of the gingival margin, indicating the extent of root surface exposure.

SECONDARY OUTCOMES:
Plaque index | Baseline
  The plaque index assesses the amount of dental plaque visible on the vestibular and lingual surfaces of all teeth
Gingival index | Baseline
  This measurement is based on the presence or absence of bleeding on gentle probing
Bleeding on probing | Baseline
  Bleeding, leading sign of inflammation inside the connective tissue, is a critical factor for pocket depth measurements, and with other variable factors prevents making reproducible measurements.
Periodontal pocket depth | Baseline
  A pathologically deepened gingival sulcus around a tooth at the gingival margin.
Clinical attachment level | Baseline
  CAL is calculated by subtracting the gingival margin level from the probing depth.

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant İzzet Baysal University, Bolu, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No